CLINICAL TRIAL: NCT00841087
Title: A 6-week, Randomised, Multi-centre, Open-labelled, Parallel Group, Exploratory Trial to Investigate the Safety of SIBA Once Daily + NovoRapid® Compared to Insulin Detemir Once Daily + NovoRapid®, All in a Basal-bolus Regimen in Subjects With Type 1 Diabetes Mellitus
Brief Title: Comparison of NN1250 Versus Insulin Detemir, Both Combined With Insulin Aspart in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3569; JapicCTI-090711 (Registry Identifier: JAPIC)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIBA (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- Insulin Detemir (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec — The insulin NN1250 (insulin degludec) injected subcutaneously at bedtime
  Arms: SIBA
Drug: insulin detemir — Injection subcutaneously at bedtime
  Arms: Insulin Detemir
Drug: insulin aspart — Injection subcutaneously immediately before each meal.

SUMMARY:
This trial is conducted in Japan. The aim of this clinical trial is to investigate the safety (with emphasis on hypoglycaemia) after switching from long-acting insulin analogue or intermediate-acting insulin to insulin degludec (NN1250, SIBA) on a basal-bolus regimen in subjects with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 1 diabetes mellitus more than one year
* Current treatment: basal (once daily at bedtime) - bolus (three times a day just before main meals) regimen only for at least 12 weeks using a long-acting insulin analogue excluding insulin detemir or intermediate-acting insulin as a basal insulin and NovoRapid® as bolus insulin (a brand of basal insulin preparation has not been changed in the preceding 12 weeks)
* HbA1c below 10.0%
* Body Mass Index (BMI) below 30.0 kg/m^2

Exclusion Criteria:

* Known hypoglycaemia unawareness or recurrent major hypoglycaemia
* Current treatment with total insulin dose of more than 100 U or IU/day
* Current treatment or expected to start treatment with systemic corticosteroid

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (7):
- Japan (7):
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Ebina-shi
  - Novo Nordisk Investigational Site, Koriyama-shi, Fukushima
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Yokohama

REFERENCES:
- [Result] Iwamoto Y, Clauson P, Nishida T, Kaku K. Insulin degludec in Japanese patients with type 1 diabetes mellitus: A randomized controlled trial. J Diabetes Investig. 2013 Jan 29;4(1):62-8. doi: 10.1111/j.2040-1124.2012.00240.x. Epub 2012 Sep 14. PMID 24843632
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 sites in Japan
Pre-assignment Details: The period between the Visit 1 (screening visit) and Visit 2 (baseline visit) of 3 weeks [±7 days] was the run-in period. The subjects continued their insulin treatment (basal-bolus therapy: insulin glargine or neutral protamine Hagedorn (intermediate-acting insulin) [NPH] insulin) same as their pre-trial dose.
Groups:
- SIBA: Soluble insulin basal analogue (SIBA, insulin degludec) was given subcutaneously once daily (OD) at bedtime and insulin aspart was given subcutaneously immediately before meals three times a day for 6 weeks. Insulin doses were individually adjusted.
- Insulin Detemir: Insulin detemir was given subcutaneously once daily (OD) at bedtime and insulin aspart was given subcutaneously immediately before meals three times a day for 6 weeks. Insulin doses were individually adjusted.
Period: Overall Study
Arm/Group | SIBA | Insulin Detemir
Started | 33 | 32
Completed | 33 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SIBA | Insulin Detemir | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (15.0) | 43.2 (15.4) | 44.4 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 24 | 19 | 43
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.39 (0.86) | 7.32 (0.86) | 7.35 (0.86)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 181.8 (66.2) | 141.8 (54.3) | 162.1 (63.4)
Body weight [Mean (Standard Deviation); unit: kg] | 64.15 (11.11) | 62.28 (7.85) | 63.23 (9.61)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Major and Minor Hypoglycaemic Episodes
Description: Observed rate of major and minor hypoglycaemic episodes per patient year (1year=365.25days) of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose ≤ 55 mg/dL.
Time Frame: Week 0 to Week 6 + 5 days follow up
Population: The Safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes /year of patient exposure
Arm/Group | SIBA | Insulin Detemir
Number analyzed (Participants) | 33 | 32
Episodes /year of patient exposure
  Major | 0 | 0
  Minor | 62.97 | 80.84

2. Primary Outcome: Rate of Nocturnal Major and Minor Hypoglycaemic Episodes
Description: Observed rate of nocturnal major and minor hypoglycaemic episodes per patient year (1year=365.25days) of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose ≤ 55 mg/dL. Episodes were defined as nocturnal if the time of onset was between 23:00-05:59 (both inclusive).
Time Frame: Week 0 to Week 6 + 5 days follow up
Population: as for outcome 1
Measure: Number; unit: Episodes /year of patient exposure
Arm/Group | SIBA | Insulin Detemir
Number analyzed (Participants) | 33 | 32
Episodes /year of patient exposure
  Major | 0 | 0
  Minor | 4.97 | 15.83

3. Secondary Outcome: Number of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to number of adverse events. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 6 + 5 days follow up
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | SIBA | Insulin Detemir
Number analyzed (Participants) | 33 | 32
events
  Adverse events (AEs) | 13 | 15
  Serious AEs | 0 | 0
  Severe AEs | 0 | 0
  Moderate AEs | 0 | 2
  Mild AEs | 13 | 13

4. Secondary Outcome: Change in Body Weight
Description: Observed change from baseline in body weight after 6 weeks of treatment
Time Frame: Week 0, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | SIBA | Insulin Detemir
Number analyzed (Participants) | 33 | 32
kg | 0.22 (1.02) | -0.20 (1.19)

5. Secondary Outcome: Electrocardiogram (ECG)
Description: The number of subjects having a electrocardiogram (ECG) that changed from 'Normal' or 'Abnormal, not clinically significant' to 'Abnormal, clinically significant'. 'Abnormal, Clinically significant' is an abnormality that suggests a disease and/or organ toxicity and is of a severity, which requires active management.
Time Frame: Week 0, Week 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SIBA | Insulin Detemir
Number analyzed (Participants) | 33 | 32
participants | 0 | 0

6. Secondary Outcome: Diastolic Blood Pressure (BP)
Description: Mean values at baseline (Week 0) and at Week 6
Time Frame: Week 0, Week 6
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIBA | Insulin Detemir
Number analyzed (Participants) | 33 | 32
mmHg
  Week 0 (Baseline) | 73.9 (7.8) | 73.8 (9.3)
  Week 6 | 74.7 (6.4) | 73.0 (8.0)

7. Secondary Outcome: Systolic Blood Pressure (BP)
Description: Mean values at baseline (Week 0) and at Week 6
Time Frame: Week 0, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIBA | Insulin Detemir
Number analyzed (Participants) | 33 | 32
mmHg
  Week 0 (Baseline) | 125.0 (15.5) | 125.3 (16.0)
  Week 6 | 125.5 (13.3) | 120.2 (13.8)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 6 weeks + 5 days follow up
Description: The Safety analysis set included all subjects who were randomised and received at least one dose of the investigational product or its comparator.
Arm/Group | SIBA | Insulin Detemir
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 5/33 | 2/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIBA (N=33) | Insulin Detemir (N=32)
Nasopharyngitis (Infections and infestations) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.